CLINICAL TRIAL: NCT02517255
Title: Salvage of Myocardial Infarction Documented by Magnetic Resonance Imaging in Patients Undergoing Rescue Percutaneous Coronary Intervention
Brief Title: Salvage of Myocardial Infarction Documented by MRI in Patients Undergoing Rescue Percutaneous Coronary Intervention
Acronym: SAVEME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luiz Fernando Ybarra, MD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 518.844
Record Dates: First submitted 2015-07-27; First posted 2015-08-06 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: ST segment elevation myocardial infarction; Failed Thrombolysis; Rescue Percutaneous Coronary Intervention; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Magnetic Resonance Imaging (Experimental): Cardiac MRI will be performed within 7 days of rescue percutaneous coronary intervention (PCI) and after 3 and 6 months.
  Interventions: Device: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Device: Cardiac Magnetic Resonance Imaging — 7 day-Cardiac MRI: T1 and T2 images; 3 and 6 month-Cardiac MRI: T1, T2 and stress perfusion images

SUMMARY:
Atherosclerotic disease is responsible for one third of all deaths annually and is a major cause of comorbidities. While atherosclerosis is by itself a benign disease, it often leads to complications such as acute myocardial infarction with ST-segment elevation. Rescue angioplasty is indicated if thrombolytic therapy fails. However, the benefits in reducing mortality and the amount of myocardium effectively saved are not well established. The development of new tools, including cardiac magnetic resonance imaging to identify myocardial area at risk and infarcted increased diagnostic accuracy. However, unlike the context of primary angioplasty, little is known about the relation between coronary epicardial and microvascular flow after rescue angioplasty and myocardial salvage. The objective of this study is to evaluate whether there is a relation between these flows and myocardial salvage identified by Magnetic Resonance Imaging (MRI). At the end of this research, the investigators hope to contribute to a better understanding of coronary flow and its relation to the amount of heart muscle saved after rescue angioplasty. This is an important information that can help understand which cases benefit most from rescue angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST segment elevation myocardial infarction (STEMI) who underwent Thrombolysis within 12 hours of chest pain and present clinical and/or electrocardiogram (EKG) signs of failed thrombolysis with indication of rescue percutaneous coronary intervention (PCI).

Exclusion Criteria:

* Patients with contraindication to Cardiac Magnetic Resonance Imaging (MRI) (pacemaker, aneurysm clip, claustrophobia, hemodynamic instability, etc).
* Allergy or contraindication to Gadolinium.
* Contraindication to dual anti-platelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Microvascular obstruction - percentage of left ventricular mass displaying a lack of contrast uptake in the core of an area showing delayed enhancement. | 6 months

SECONDARY OUTCOMES:
Infarct size - percentage of left ventricular mass with signal intensity 2 standard deviations above the mean signal obtained in the remote non-infarcted myocardium. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Carvalho, MD, PhD, Study Chair — Full Professor at Universidade Federal de São Paulo
Locations (1):
- Escola Paulista de Medicina - Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil